CLINICAL TRIAL: NCT04448262
Title: Bronchial Asthma and Diabetes: Impact on Bronchial Inflammation and Exercise Capacity
Status: Terminated | Type: Observational
Why Stopped: technical issue
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: Galmarini Hospital, Tradate (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2290 CE
Record Dates: First submitted 2020-04-07; First posted 2020-06-25 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Asthma; Diabete Type 2
Keywords: eosinophils, symptoms, lung
MeSH Terms: conditions — Asthma; Diabetes Mellitus, Type 2 | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- G1 Asthma: Diagnosis of bronchial asthma according to the Global Initiative for Asthma (GINA) 2018 guideline Clinical stability of asthmatic disease Age ≥18 years Not-smokers, smokers or ex-smokers with pack/year ≤10
  Interventions: Other: data collection
- G2 Diabetes: Diagnosis of Type II diabetes according to the last Italian guidelines and HbA1c < 9%, 54-75mmol/mol Age ≥18 years Not-smokers, smokers or ex-smokers with pack/year ≤10
  Interventions: Other: data collection
- G3 Asthma plus diabetes: Concomitant diagnosis of bronchial asthma according to the GINA 2018 guideline, Clinical stability of asthmatic disease and Diagnosis of Type II diabetes according to the last Italian guidelines and HbA1c < 9%, 54-75mmol/mol Age ≥18 years Not-smokers, smokers or ex-smokers with pack/year ≤10
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — collection of data about bronchial and systemic inflammation, quality of life, lung function

SUMMARY:
Type 2 diabetes is the most common form of diabetes and according to several studies, even lung can represent another target of the diabetic disease. Asthmatic patients often show comorbidities and obesity is one of the main.Several studies in literature suggest that patients with higher Body Mass Index (i.e. overweight and obese) have a greater risk of developing asthma compared to normal weight subjects. Considering inflammation, asthma is usually characterized by an increase of eosinophils in the airways and by a Th2 type inflammation, while a immunological type Th1 switch systemically characterizes diabetes. Even asthmatic patients, especially if diabetic, might have an increase of glucose in their airways, that could favourite or feed an inflammatory/infective state. Up to-day there are not in literature studies that have investigated the airways inflammatory pattern and the exercise capacity in relation to functional characteristics in diabetic patients affected by asthma.

DETAILED DESCRIPTION:
The basic therapy for asthma treatment involves the use of corticosteroids that can lead to the development of glucose intolerance and to the onset of diabetes. Moreover, several works in literature highlight the fact that patients with diagnosis of both asthma and diabetes have a scarcer glycaemic control, a reduced life expectancy, and a higher risk of pneumonia when compared to patients with only asthma or only diabetes.

However, in the last years the evaluation of the inflammatory patterns in asthmatic patients has revealed a heterogeneity of the inflammation, with patients characterized by neutrophilic phenotype, mixed granulocytic or without a well-defined inflammatory component (pauci-granulocytic phenotype).On the other side, a immunological type Th1 switch systemically characterizes diabetes. The impact of diabetes, therefore, as a comorbidity in asthmatic patients could influence the inflammatory status of airways. Moreover, studies have reported that glucose is higher in the airways of subjects affected by chronic obstructive pulmonary disease and it correlates with bacterial and viral load compared to healthy controls. Even asthmatic patients, especially if diabetic, might have an increase of glucose in their airways, that could favourite or feed an inflammatory/infective state. Although physical exercise is able to reduce the level of systemic inflammation, improving asthma symptoms and glycaemic control, it is well known that asthmatic and diabetic patients tend to lead a more sedentary life style compared to healthy subjects.A limiting factor that bonds the two pathologies is obesity, since the gain of weight causes exacerbation of respiratory symptoms, resulting in lower effort tolerance.

Up to-day there are not in literature studies that have investigated the airways inflammatory pattern and the exercise capacity in relation to functional characteristics in diabetic patients affected by asthma.

Aim of the study is to characterize the airways inflammatory pattern of patients affected by bronchial asthma, patients affected by type II diabetes and patients with concomitant diagnosis of asthma and diabetes by using induced sputum. Secondary objective is to characterize the exercise capacity in relation to the functional and anthropometric characteristics of patients with diabetes, with asthma and diabetes, compared to patients with only asthma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bronchial asthma according to the GINA 2018 guideline
* Clinical stability of asthmatic disease
* Diagnosis of Type II diabetes according to the last Italian guidelines (1) and HbA1c < 9%, 54-75mmol/mol
* Concomitant diagnosis of bronchial asthma (12) and diabetes according to the described guidelines
* Age ≥18 years
* Not-smokers, smokers or ex-smokers with pack/year ≤10
* Patients able to collaborate in the required procedures and who have signed the informed consent

Exclusion criteria:

* Bronchial asthma and/or diabetes with scarce clinical control.
* Diagnosis of cognitive impairment
* Not able to carry out study procedures

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthmatic patients will be evaluated and enrolled during outpatients follow-up visits at the ICS Institute Maugeri of Tradate, type II diabetic patients at the Galmarini Hospital of Tradate, while patients with concomitant diagnosis of asthma and type II diabetes will be evaluated and enrolled and enrolled in both the two structures.
  20 patients per group will be the sample size
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
inflammatory cells | baseline
  macrophages%,neutrophils%, eosinophils%, lymphocytes%

SECONDARY OUTCOMES:
Expiratory muscles strength | baseline
  Maximal inspiratory pressure -MIP, Maximal expiratory pressure -MEP
Functional capacity of exercise | baseline
  6 minutes walking test-6MWT
Dyspnoea and muscular fatigue | baseline
  Dyspnoea and muscle fatigue measured with Modified Borg Scale (0-10, where 0 is better)
peripheral muscle strength | baseline
  Five Sit to Stand Test-5STS
Health related Quality of life | baseline
  St. George Respiratory Questionnaire-SGRQ, scores range from 0 to 100, with higher scores indicating more limitations
perceived Health state | baseline
  Chronic Obstructive Pulmonary Disease Assessment test-CAT, Scores range from 0 to 40, with higher scores indicating worse health state

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Spanevello, Prof, Study Director — ICS Maugeri
Locations (1):
- Istituti Clinici Maugeri Pneumologia, Tradate, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vracko R, Thorning D, Huang TW. Basal lamina of alveolar epithelium and capillaries: quantitative changes with aging and in diabetes mellitus. Am Rev Respir Dis. 1979 Nov;120(5):973-83. doi: 10.1164/arrd.1979.120.5.973. PMID 507532
- [Background] Visca D, Pignatti P, Spanevello A, Lucini E, La Rocca E. Relationship between diabetes and respiratory diseases-Clinical and therapeutic aspects. Pharmacol Res. 2018 Nov;137:230-235. doi: 10.1016/j.phrs.2018.10.008. Epub 2018 Oct 9. PMID 30312663
- [Background] Cardet JC, Ash S, Kusa T, Camargo CA Jr, Israel E. Insulin resistance modifies the association between obesity and current asthma in adults. Eur Respir J. 2016 Aug;48(2):403-10. doi: 10.1183/13993003.00246-2016. Epub 2016 Apr 21. PMID 27103388
- [Background] Mallia P, Webber J, Gill SK, Trujillo-Torralbo MB, Calderazzo MA, Finney L, Bakhsoliani E, Farne H, Singanayagam A, Footitt J, Hewitt R, Kebadze T, Aniscenko J, Padmanaban V, Molyneaux PL, Adcock IM, Barnes PJ, Ito K, Elkin SL, Kon OM, Cookson WO, Moffat MF, Johnston SL, Tregoning JS. Role of airway glucose in bacterial infections in patients with chronic obstructive pulmonary disease. J Allergy Clin Immunol. 2018 Sep;142(3):815-823.e6. doi: 10.1016/j.jaci.2017.10.017. Epub 2018 Jan 5. PMID 29310905